CLINICAL TRIAL: NCT02950051
Title: A Phase 3 Multicenter, Randomized, Prospective, Open-label Trial of Standard Chemoimmunotherapy (FCR/BR) Versus Rituximab Plus Venetoclax (RVe) Versus Obinutuzumab (GA101) Plus Venetoclax (GVe) Versus Obinutuzumab Plus Ibrutinib Plus Venetoclax (GIVe) in Fit Patients with Previously Untreated Chronic Lymphocytic Leukemia (CLL) Without Del(17p) or TP53 Mutation
Brief Title: Standard Chemoimmunotherapy (FCR/BR) Versus Rituximab + Venetoclax (RVe) Versus Obinutuzumab (GA101) + Venetoclax (GVe) Versus Obinutuzumab + Ibrutinib + Venetoclax (GIVe) in Fit Patients with Previously Untreated Chronic Lymphocytic Leukemia (CLL) Without Del(17p) or TP53 Mutation
Acronym: GAIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); Hoffmann-La Roche (Industry); AbbVie (Industry); Stichting Hemato-Oncologie voor Volwassenen Nederland (Other); Nordic CLL Study Group (NCLLSG) (Unknown); Swiss Cancer Institute (Other); Cancer Trials Ireland (Network); Israeli CLL Study Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL13; 2015-004936-36 (EudraCT Number)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2024-12-30 (Actual); Status verified 2024-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Cyclophosphamide; Rituximab; Bendamustine Hydrochloride; venetoclax; obinutuzumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard chemoimmunotherapy (SCIT) (Active Comparator): Patients up to age 65: 6 cycles (q28d) of Fludarabine + Cyclophosphamide + Rituximab (FCR)
  Patients older than 65 years: 6 cycles (q28d) of Bendamustine + Rituximab (BR)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: Rituximab; Drug: Bendamustine
- Rituximab + Venetoclax (RVe) (Experimental): 6 cycles (q28d) of RVe + 6 cycles (q28d) of Venetoclax (alone)
  Interventions: Biological: Rituximab; Drug: Venetoclax
- Obinutuzumab + Venetoclax (GVe) (Experimental): 6 cycles (q28d) of GVe + 6 cycles (q28d) of Venetoclax (alone)
  Interventions: Drug: Venetoclax; Biological: Obinutuzumab
- Obinutuzumab + Ibrutinib + Venetoclax (GIVe) (Experimental): 6 cycles (q28d) of GIVe + 6 cycles (q28d) of Ibrutinib plus Venetoclax.
  Administration of ibrutinib will be continued for a maximum of 36 months or until MRD negativity, start of new anti-CLL therapy or inacceptable toxicity, whatever occurs first.
  Interventions: Drug: Venetoclax; Biological: Obinutuzumab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Fludarabine — Fludarabine i.v.: cycles 1-6: 25 mg/m², d1-3, q28d
  Other Names: Fludura
  Arms: Standard chemoimmunotherapy (SCIT)
Drug: Cyclophosphamide — Cyclophosphamide i.v.: cycles 1-6: 250 mg/m², d1-3, q28d
  Other Names: Endoxan
  Arms: Standard chemoimmunotherapy (SCIT)
Biological: Rituximab — Rituximab i.v. (before chemotherapy): cycle 1: 375 mg/m², d0; cycles 2-6: 500 mg/m², d1; q28d
  Other Names: MabThera; Rituxan
  Arms: Rituximab + Venetoclax (RVe); Standard chemoimmunotherapy (SCIT)
Drug: Bendamustine — Bendamustine i.v.: cycles 1-6: 90mg/m², d1-2, q28d
  Other Names: Ribomustin; Levact
  Arms: Standard chemoimmunotherapy (SCIT)
Drug: Venetoclax — Venetoclax p.o. (ramp-up: dose escalation until final dose is reached)
  cycle 1: 20 mg (2 tabl. at 10 mg), d22-28, q28d
  cycle 2: 50 mg (1 tabl. at 50 mg), d1-7; 100 mg (1 tabl. at 100 mg), d8-14; 200 mg (2 tabl. at 100 mg), d15-21; 400 mg (4 tabl. at 100 mg), d22-28, q28d
  cycles 3-12: 400 mg (4 tabl. at 100 mg), d1-28, q28d
  Other Names: Venclexta; Venclyxto
  Arms: Obinutuzumab + Ibrutinib + Venetoclax (GIVe); Obinutuzumab + Venetoclax (GVe); Rituximab + Venetoclax (RVe)
Biological: Obinutuzumab — Obinutuzumab i.v.
  cycle 1: 100 mg, d1; 900 mg, d1(2); 1000 mg, d8+15, q28d
  cycles 2-6: 1000 mg, d1, q28d
  Other Names: Gazyva; Gazyvaro
  Arms: Obinutuzumab + Ibrutinib + Venetoclax (GIVe); Obinutuzumab + Venetoclax (GVe)
Drug: Ibrutinib — Ibrutinib p.o.
  cycles 1-12: 420 mg, d1-28, q28d
  cycles 13-36: 420 mg, d1-28, q28d
  Other Names: Imbruvica
  Arms: Obinutuzumab + Ibrutinib + Venetoclax (GIVe)

SUMMARY:
The aim of this study is to evaluate if standard chemoimmunotherapy (FCR, BR) in frontline treatment of physically fit CLL patients without del17p or TP 53 mutation can be replaced by combinations of targeted drugs (Venetoclax, Ibrutinib) with anti-CD20-antibodies (Rituximab, Obinutuzumab), which may induce extremely long lasting remissions.

DETAILED DESCRIPTION:
Chemoimmunotherapy is the standard of care in first-line treatment of CLL patients without del17p or TP 53 mutation; physically fit patients are treated with fludarabine, cyclophosphamide and rituximab (FCR)1. Due to the high risk of severe neutropenias and infections with FCR, bendamustine and rituximab (BR) must be considered in patients aged >65 years.

However, these conventional chemoimmunotherapies are associated with side effects caused by the rather unspecific mode of action of the chemotherapy. Therefore, there is an urgent need for alternatives, especially chemotherapy-free regimens.

In first line treatment of elderly patients with CLL and coexisting conditions, the anti-CD20-antibody obinutuzumab is the new standard therapy. In the CLL11 trial the combination of obinutuzumab with chlorambucil proved to be safe and lead to markedly improved response rates as well as PFS times in comparison to chlorambucil alone or combined with rituximab.

The BCL2 antagonist venetoclax (GDC-0199/ABT-199) showed striking activity with tumor lysis syndrome as dose limiting toxicity in patients with relapsed and refractory CLL. 400 mg venetoclax was determined to be a safe and efficacious dose. Several patients treated with the combination of venetoclax and rituximab in relapsed refractory CLL even achieved MRD negativity. The FDA approved Venetoclax for the treatment of relapsed CLL with 17p/TP53 on 12th April 2016.

Therefore, venetoclax plus CD20-antibody based combinations have the potential to induce higher rates of MRD negativity in frontline therapy of CLL and concomitantly induce lower rates of toxicities so that chemotherapy might be replaced. Furthermore, venetoclax and obinutuzumab demonstrated synergistic activity in a preclinical study of a murine Non-Hodgkin lymphoma xenograft model, and additive activity in a CLL lymph node model. The combination appears tolerable in the firstline treatment of CLL patients with coexisting conditions whilst the toxicity profile of both drugs compares favorably to those of the chemotherapies currently used in the treatment of CLL. Consequently, it should be tested if rituximab can be replaced by obinutuzumab in combination with venetoclax in this trial.

Ibrutinib, a selective, irreversible small molecular inhibitor of Bruton´s Tyrosine Kinase (BTK), showed excellent responses and a safe toxicity profile9,10, even in combination with BR. Ibrutinib is approved for treatment of relapsed CLL as well as frontline therapy of CLL by the FDA and EMA (April 29th 2016).

The combination of ibrutinib and venetoclax showed synergy in primary CLL cells.

Consequently, the aim of the current trial is to evaluate if chemoimmunotherapy in the frontline treatment of physically fit patients in CLL can be replaced by combinations of these targeted drugs with anti-CD20-antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Documented CLL requiring treatment according to iwCLL criteria
2. Age at least 18 years
3. Life expectancy ≥ 6 months
4. Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements
5. Adequate bone marrow function indicated by a platelet count >30 x10^9/l (unless directly attributable to CLL infiltration of the bone marrow, proven by bone marrow biopsy)
6. Creatinine clearance ≥70ml/min directly measured with 24hr urine collection or calculated according to the modified formula of Cockcroft and Gault (for men: GFR ≈ ((140 - age) x bodyweight) / (72 x creatinine), for women x 0, 85). For patients with creatinine values within the normal range the calculation of the clearance is not necessary. Dehydrated patients with an estimated creatinine clearance less than 70 ml/min may be eligible if a repeat estimate after adequate hydration is > 70 ml/min
7. Adequate liver function as indicated by a total bilirubin≤ 2 x, AST/ALT ≤ 2.5 x the institutional ULN value, unless directly attributable to the patient's CLL or to Gilbert's Syndrome
8. Negative serological testing for hepatitis B (HBsAg negative and anti-HBc negative; patients positive for anti-HBc may be included if PCR for HBV DNA is negative and HBV-DNA PCR is performed every month until 12 months after last treatment cycle), negative testing for hepatitis C RNA within 6 weeks prior to registration
9. Eastern Cooperative Oncology Group Performance Status (ECOG) performance status 0-2

Exclusion Criteria:

1. Any prior CLL-specific therapies (except corticosteroid treatment administere due to necessary immediate intervention; within the last 10 days before start of study treatment, only dose equivalents of 20 mg prednisolone are permitted).
2. Transformation of CLL (Richter transformation)
3. Decompensated hemolysis, defined as ongoing hemoglobin drop in spite of three more concurrent treatments being administered for hemolysis
4. Detected del(17p) or TP53 mutation
5. Patients with a history of PML
6. Any comorbidity or organ system impairment rated with a single CIRS (cumulative illness rating scale) score of 4 (excluding the eyes/ears/nose/throat/larynx organ system), a total CIRS score of more than 6 or any other life-threatening illness, medical condition or organ system dysfunction that, in the investigator´s opinion, could comprise the patients safety or interfere with the absorption or metabolism of the study drugs (e.g, inability to swallow tablets or impaired resorption in the gastrointestinal tract)
7. Urinary outflow obstruction
8. Malignancies other than CLL currently requiring systemic therapies, not being treated in curative intention before (unless the malignant disease is in a stable remission due to the discretion of the treating physician) or showing signs of progression after curative treatment
9. Uncontrolled or active infection
10. Patients with known infection with human immunodeficiency virus (HIV)
11. Requirement of therapy with strong CYP3A4 and CYP3A5 inhibitors/inducers
12. Anticoagulant therapy with warfarin or phenoprocoumon, (rotation to alternative anticoagulation is allowed, but note that patients being treated with NOAKs can be included, but must be properly informed about the potential risk of bleeding under treatment with ibrutinib)
13. History of stroke or intracranial hemorrhage within 6 months prior to registration
14. Use of investigational agents which might interfere with the study drug within 28 days prior to registration
15. Vaccination with live vaccines 28 days prior to registration
16. Major surgery less than 30 days before start of treatment
17. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, known sensitivity or allergy to murine products
18. Known hypersensitivity to any active substance or to any of the excipients of one of the drugs used in the trial
19. Pregnant women and nursing mothers (a negative pregnancy test is required for all women of childbearing potential within 7 days before start of treatment; further pregnancy testing will be performed regularly)
20. Fertile men or women of childbearing potential unless:

    1. surgically sterile or ≥ 2 years after the onset of menopause
    2. willing to use two methods of reliable contraception including one highly effective contraceptive method (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 18 months after the end of study treatment
21. Legal incapacity
22. Prisoners or subjects who are institutionalized by regulatory or court order
23. Persons who are in dependence to the sponsor or an investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 926 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Miminimal residual disease (MRD) negativity rate in peripheral blood (PB) | Month 15
  Proportion of MRD negative patients at month15 based on the intention-to-treat population (ITT population), that is the number of MRD negative patients divided by the number of the ITT population. MRD negativity is defined as <1 CLL-cell among 10,000 leukocytes analyzed [0.01%], i.e. < 10-4.
  Primary outcome measure for the comparison of GVe vs. SCIT
Progression free survival (PFS) | anticipated for January 2023 (after 213 events occured and 73 months after the first patient has been randomized
  Time from randomization to the first occurrence of progression or relapse (determined using standard IWCLL guidelines [2008]), or death from any cause, whichever occurs first.
  Primary outcome measure for the comparison GIVe vs. SCIT

SECONDARY OUTCOMES:
MRD negativity rate in PB | Month 15
  Time from randomization to the first occurrence of progression or relapse (determined using standard IWCLL guidelines [2008]), or death from any cause, whichever occurs first.
  Secondary outcome measure for all other comparisons with the exception of GVe vs. SCIT
MRD levels in PB | Month 2, 9, 13 and later time points according to the discretion of the treating physician at local laboratories
MRD levels in bone marrow (BM) | at final restaging (RE): 2 month after the end of the last treatment cycle
PFS | anticipated for January 2023 (after 213 events occured and 73 months after the first patient has been randomized)
  Time from randomization to the first occurrence of progression or relapse (determined using standard IWCLL guidelines [2008]), or death from any cause, whichever occurs first.
  Secondary outcome measure for all other comparisons with the exception of GIVe vs.SCIT
Overall response rate (ORR) | Month 3, 9, 13 and 15
Rate of complete responses (CR) / complete responses with incomplete bone marrow recovery(CRi) | Interim staging (IST: cycle 4 d1), cycle 9 d1 (or final restaging (RE) for patients in the SCIT arm), IR (or three month after RE for patients in the SCIT arm respectively) and Month 15, with regard to best response achieved
  Complete response (CR) rate is defined by the proportion of patients having achieved a CR/CRi defined by the IWCLL guidelines as best response until and including the response assessment at Month 6, 9, 12 and 15 (= number of patients with best response CR/CRi divided by the ITT population).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Eichhorst, MD, Prof., Principal Investigator — Department I of Internal Medicine, University Hospital Cologne
Locations (161):
- Austria (3):
  - Medizinische Universitaet Wien, Vienna
  - Hanusch Hospital, Vienna
  - Wilhelminenspital, Vienna
- Belgium (5):
  - ZNA Stuivenberg, Antwerp
  - Algemeen Ziekenhuis St. Jan, Bruges
  - Jan Yperman Ziekenhuis, Ieper
  - UZ Gasthuisberg, Leuven
  - AZ Delta, Roeselare
- Denmark (9):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet/Copenhagen, Copenhagen
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - University Hospital Herlev, Herlev
  - Regionshospitalet Holstebro, Holstebro
  - Odense Universitets Hospital, Odense
  - Sjællands Universitetshospital, Roskilde
  - Vejle Hospital, Vejle
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Jyväskylä Central Hospital, Jyväskylä
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Germany (70):
  - Gesundheitszentrum Klinikum St Marien, Amberg
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Helios-Klinikum Berlin, Berlin
  - ZAHO Bonn, Bonn
  - Ev. Diakonie-Krankenhaus gemeinnuetzige GmbH, Bremen
  - University Hospital of Cologne, Cologne
  - St. -Johannes-Hospital Dortmund, Dortmund
  - Gefos Dortmund mbH, Dortmund
  - BAG Dresden, Dresden
  - Universitaetsklinik Carl Gustav Carus, Dresden
  - Marien Hospital Düsseldorf GmbH, Düsseldorf
  - St. Georg Klinikum Eisenach GmbH, Eisenach
  - Helios Klinikum Erfurt, Erfurt
  - St. Antonius-Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Centrum fuer Haematologie und Onkologie Bethanien, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - MVZ Onkologische Kooperation Harz, Drs. Tessen/Hoyer/Zahn, Goslar
  - Onkologische Schwerpunktpraxis Göttingen, Göttingen
  - Universitaetsmedizin Göttingen, Göttingen
  - Universitaetsmedizin Greifswald, Greifswald
  - UKE Hamburg, Hamburg
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - EVK Hamm, Hamm
  - MediProjekt GBR, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Marienhospital Herne, Herne
  - Onkologische Schwerpunktpraxis Des. Freier/Sievers, Hildesheim, Hildesheim
  - Universitaetsklinikum Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Städt. Klinikum Karlsruhe, Karlsruhe
  - Dres. Siehl / Soeling, Fachaerzte fuer Haematologie und Internistische Onkologie, Kassel, Kassel
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - InVO-Institut fuer Versorgungsforschung in der Onkologie GbR, Koblenz
  - Tagesklinik Landshut, Dr. Vehling-Kaiser, Landshut
  - Gemeinschaftspraxis Haemato/ Onkologie Lebach, Lebach
  - Onkologische Schwerpunktpraxis Dr. Mueller, Leer, Leer
  - Klinikum Lippe GmbH, Lemgo
  - Gemeinschaftspraxis Haematologie und Onkologie, Magdeburg
  - Universitaetsklinikum Magdeburg, Magdeburg
  - Universitaetsklinik Mainz, Mainz
  - Mannheimer Onkologie Praxis, Mannheim
  - Institut fuer Versorgungsforschung Dr. med. M. Maasberger/ M. Schmitz/ Dr. med. M. T. Keller, Mayen
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Stauferklinikum Schwaebisch-Gmuend, Mutlangen
  - MVZ MOP Elisenhof, München
  - Klinikum Schwabing, München
  - Ludwig-Maximilians-Universitaet Muenchen, München
  - Klinikum rechts der Isar, München
  - Haematologische/Onkologische Praxis Neunkirchen, Neunkirchen
  - Studiengesellschaft Onkologie Rhein Ruhr, Oberhausen
  - Gemeinschaftspraxis Dres. Ballo/Boeck, Offenbach
  - Klinik fuer Haematologie und Onkologie, Paderborn
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Krankenhaus der Barmherzigen Brüder, Regensburg
  - OncoPro GbR, Regensburg
  - Universitätsmedizin Rostock, Rostock
  - Praxis für Hämatologie und Onkologie Dres. Jacobs/Daus/Schmits, Saarbrücken
  - Leopoldina-Krankenhaus, Schweinfurt
  - ZAHO-Rheinland, Siegburg
  - Marienhospital Stuttgart, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - MVZ Weiden GmbH, Weiden
  - Haematologisch-Onkologische Schwerpunktpraxis Dres. Perker/Sandherr, Weilheim, Weilheim
  - Helios Klinikum Wuppertal, Wuppertal
  - Gemeinschaftspraxis Dr. Schlag/Dr. Schoettker, Würzburg
  - Universitaetsklinik Wuerzburg, Würzburg
- Ireland (6):
  - Cork University Hospital, Cork
  - Mater Misericordiae Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Waterford, Waterford
- Israel (6):
  - Bnai-Zion Medical. Il-Haifa, Haifa
  - Hadassah Ein Kerem, Jerusalem
  - Meir Medicail Center, Kfar Saba
  - Rabin medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Souraski Tel-Aviv Medical Center, Tel Aviv
- Netherlands (33):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - MC Alkmaar, Alkmaar
  - Meander Medisch Centrum, Amersfoort, Amersfoort
  - VUmc, Amsterdam, Amsterdam
  - NL-Amsterdam-AMC, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - Amphia Ziekenhuis, Breda
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Reinier de Graaf Gasthuis, Delft
  - Deventer ziekenhuizen, Deventer
  - Albert Schweitzer Ziekenhuis, Dordrecht, Dordrecht
  - Gelderse Vallei, Ede
  - Maxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Groene Hart Ziekenhuis, Gouda
  - UMCG, Groningen
  - Ziekenhuisgroep Twente Hengelo, Hengelo
  - Tergooi Ziekenhuis, Hilversum
  - Spaarne Ziekenhuis, Hoofddorp
  - Medisch Centrum Leeuwarden Zuid, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht university medial Center, Maastricht
  - St. Antonius Ziekehuis, Nieuwegein
  - Radboud UMC, Nijmegen
  - Canisius-Wilhelmina ZH, Nijmegen
  - Maasstadziekenhuis, Rotterdam
  - Antonius Ziekenhuis Sneek, Sneek
  - ZorgSaam Zeeuws Vlaanderen, Terneuzen
  - St. Elisabeth ZH, Tilburg
  - UMCU, Utrecht
  - VieCuri loc. Venlo, Venlo
  - Zaans Medisch Centrum, Zaandam
  - Isala, Zwolle
- Sweden (9):
  - Soedra Aelvsborgs Sjukhus, Borås
  - Falu lasarett, Falun
  - Hallands hospital - Halmstad, Halmstad
  - Universitetsjukhuset i Linkoeping, Linköping
  - Sunderby Hospital, Luleå
  - Skane University Hospital Lund, Lund
  - Universitetssjukhuset i Oerebro, Örebro
  - Akademiska Sjukhuset, Uppsala
  - Hallands hospital - Varberg, Varberg
- Switzerland (15):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - IOSI, Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubunden, Chur
  - Universitaire de Geneve, Geneva
  - KSBL Liestal, Liestal
  - Luzerner Kantonsspital, Lucerne
  - Spital Thurgau AG, Münsterlingen
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - KS Winterthur, Winterthur
  - Stadtspital Triemli, Zurich
  - Universitaetsspital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furstenau M, Kater AP, Robrecht S, von Tresckow J, Zhang C, Gregor M, Thornton P, Staber PB, Tadmor T, Lindstrom V, Juliusson G, Janssens A, Levin MD, da Cunha-Bang C, Schneider C, Goldschmidt N, Vandenberghe E, Rossi D, Benz R, Nosslinger T, Heintel D, Poulsen CB, Christiansen I, Frederiksen H, Enggaard L, Posthuma EFM, Issa DE, Visser HPJ, Bellido M, Kutsch N, Durig J, Stehle A, Vohringer M, Bottcher S, Schulte C, Simon F, Fink AM, Fischer K, Holmes EE, Kreuzer KA, Ritgen M, Bruggemann M, Tausch E, Stilgenbauer S, Hallek M, Niemann CU, Eichhorst B. First-line venetoclax combinations versus chemoimmunotherapy in fit patients with chronic lymphocytic leukaemia (GAIA/CLL13): 4-year follow-up from a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2024 Jun;25(6):744-759. doi: 10.1016/S1470-2045(24)00196-7. PMID 38821083
- [Background] Eichhorst B, Niemann CU, Kater AP, Furstenau M, von Tresckow J, Zhang C, Robrecht S, Gregor M, Juliusson G, Thornton P, Staber PB, Tadmor T, Lindstrom V, da Cunha-Bang C, Schneider C, Poulsen CB, Illmer T, Schottker B, Nosslinger T, Janssens A, Christiansen I, Baumann M, Frederiksen H, van der Klift M, Jager U, Leys MBL, Hoogendoorn M, Lotfi K, Hebart H, Gaska T, Koene H, Enggaard L, Goede J, Regelink JC, Widmer A, Simon F, De Silva N, Fink AM, Bahlo J, Fischer K, Wendtner CM, Kreuzer KA, Ritgen M, Bruggemann M, Tausch E, Levin MD, van Oers M, Geisler C, Stilgenbauer S, Hallek M; GCLLSG, the HOVON and Nordic CLL Study Groups, the SAKK, the Israeli CLL Association, and Cancer Trials Ireland. First-Line Venetoclax Combinations in Chronic Lymphocytic Leukemia. N Engl J Med. 2023 May 11;388(19):1739-1754. doi: 10.1056/NEJMoa2213093. PMID 37163621
- [Derived] Langerbeins P, Giza A, Robrecht S, Cramer P, von Tresckow J, Al-Sawaf O, Fink AM, Furstenau M, Kutsch N, Simon F, Goede V, Hoechstetter M, Niemann CU, da Cunha-Bang C, Kater A, Dubois J, Gregor M, Staber PB, Tausch E, Schneider C, Stilgenbauer S, Eichhorst B, Fischer K, Hallek M. Reassessing the chronic lymphocytic leukemia International Prognostic Index in the era of targeted therapies. Blood. 2024 Jun 20;143(25):2588-2598. doi: 10.1182/blood.2023022564. PMID 38620092
- [Derived] Furstenau M, Thus YJ, Robrecht S, Mellink CHM, van der Kevie-Kersemaekers AM, Dubois J, von Tresckow J, Patz M, Gregor M, Thornton P, Staber PB, Tadmor T, Levin MD, da Cunha-Bang C, Schneider C, Poulsen CB, Illmer T, Schottker B, Janssens A, Christiansen I, Nosslinger T, Baumann M, Hebart H, Gaska T, Regelink JC, Dompeling EC, Lindstrom V, Juliusson G, Widmer A, Goede J, Goldschmidt N, Simon F, De Silva N, Fink AM, Fischer K, Wendtner CM, Ritgen M, Bruggemann M, Tausch E, Spaargaren M, Eldering E, Stilgenbauer S, Niemann CU, Hallek M, Eichhorst B, Kreuzer KA, Kater AP. High karyotypic complexity is an independent prognostic factor in patients with CLL treated with venetoclax combinations. Blood. 2023 Aug 3;142(5):446-459. doi: 10.1182/blood.2023019634. PMID 37172204
- [Derived] Furstenau M, Langerbeins P, De Silva N, Fink AM, Robrecht S, von Tresckow J, Simon F, Hohloch K, Droogendijk J, van der Klift M, van der Spek E, Illmer T, Schottker B, Fischer K, Wendtner CM, Tausch E, Stilgenbauer S, Niemann CU, Gregor M, Kater AP, Hallek M, Eichhorst B. COVID-19 among fit patients with CLL treated with venetoclax-based combinations. Leukemia. 2020 Aug;34(8):2225-2229. doi: 10.1038/s41375-020-0941-7. Epub 2020 Jun 29. No abstract available. PMID 32601378
- See also: Click here for more information about this study: CLL13 (German CLL Study Group) — https://www.dcllsg.com/cll13/